CLINICAL TRIAL: NCT06112340
Title: A Multicenter, Extension Study to Evaluate the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of Two Doses of Linsitinib in Subjects With Active, Moderate to Severe Thyroid Eye Disease (TED)
Brief Title: Extension Study of Two Doses of Linsitinib in Subjects With Active, Moderate to Severe Thyroid Eye Disease (TED)
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sling Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VGN-TED-302
Record Dates: First submitted 2023-10-16; First posted 2023-11-01 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Thyroid Eye Disease; Graves Orbitopathy; Endocrine System Diseases; Eye Diseases; Thyroid Associated Ophthalmopathy; Graves Ophthalmopathy; Thyroid Diseases; Orbital Diseases; Proptosis; IGF1R; Exophthalmos; Hashimoto
MeSH Terms: conditions — Graves Ophthalmopathy; Endocrine System Diseases; Eye Diseases; Thyroid Diseases; Orbital Diseases; Exophthalmos; Hashimoto Disease | interventions — 3-(8-amino-1-(2-phenylquinolin-7-yl)imidazo(1,5-a)pyrazin-3-yl)-1-methylcyclobutanol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Low Dose (Active Comparator): Active Arm Low Dose Linsitinib
  Interventions: Drug: linsitinib
- High Dose (Active Comparator): Active Arm High Dose Linsitinib
  Interventions: Drug: linsitinib

INTERVENTIONS:
Drug: linsitinib — Study medication taken twice daily by mouth

SUMMARY:
The overall study objective is to continue to assess the efficacy, safety, pharmacokinetics, and pharmacodynamics of linsitinib in subjects who were enrolled in the prior VGN-TED-301 through Week 24. These subjects include VGN-TED-301 Week 24 proptosis non-responders or subjects who relapse during the Follow-Up Period of VGN-TED-301.

ELIGIBILITY:
Inclusion Criteria:

* Subject who completed the 24-week double-mask period of VGN-TED-301 and are proptosis non-responders (< 2 mm reduction in proptosis in the study eye) at Week 24 of VGN-TED-301 study or proptosis responders at Week 24 who relapse during the Follow-Up period of VGN-TED-301
* Subject has not received any treatment for TED since Week 24 of VGN-TED-301
* Subjects must be euthyroid with the participant's baseline disease under control or have mild hypo- or hyperthyroidism (defined as free thyroxine [FT4] and free triiodothyronine levels [FT3] <50% above or below the normal limits) at Baseline. Every effort should be made to correct mild hypo- or hyperthyroidism promptly and maintain the euthyroid state for the duration of the clinical trial
* Does not require immediate ophthalmic surgery, radiotherapy to orbits or other ophthalmological intervention at the time of Baseline and is not planning for any such treatment during the course of the study

Exclusion Criteria:

* The exclusion criteria of protocol VGN-TED-301 also apply to this extension study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-10-11 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of Subjects who are Proptosis Responders at Week 24 | 24 weeks
  Percentage of subjects with a ≥ 2 mm reduction of proptosis from baseline as determined by exophthalmometer

SECONDARY OUTCOMES:
Change from Baseline in Proptosis to Week 24 (Study Eye) | 24 weeks
  Change from baseline in reduction of proptosis from baseline as determined by exophthalmometer
Percentage of Subjects who are Overall Responders at Week 24 | 24 weeks
  Percentage of Subjects with a response of ≥ 2 mm reduction of proptosis at Week 24 as determined by exophthalmometer
Percentage of Subjects who are CAS Categorical Responders at Week 24 (Study Eye) | 24 weeks
Change from Baseline in the Graves' Ophthalmopathy Quality of Life (GO-QoL) Questionnaire Overall Score to Week 24 | 24 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Bascom Palmer Eye Institute, Miami, Florida
  - West Virginia University Eye Institute, Morgantown, West Virginia